CLINICAL TRIAL: NCT06141096
Title: A Multi-center, Open-label, Randomized Phase II Clinical Study to Evaluate the Efficacy and Safety of I.V.Infusion of MB07133 in Patients With Unresectable HCC
Brief Title: MB07133 for the Treatment of Patients With Unresectable Hepatocellular Carcinoma
Acronym: MB07133
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H201110LC2
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Safety Issues; Effect of Drug; Tolerance
MeSH Terms: interventions — 4-amino-1-(5-O-(2-oxo-4-(4-pyridyl)-1,3,2-dioxaphosphorinan-2-yl)arabinofuranosyl)-2(1H)-pyrimidinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MB07133 600mg/m2/day (Experimental)
  Interventions: Drug: MB07133
- MB07133 1200mg/m2/day (Experimental)
  Interventions: Drug: MB07133
- MB07133 1800mg/m2/day (Experimental)
  Interventions: Drug: MB07133

INTERVENTIONS:
Drug: MB07133 — Evaluate the effectiveness and safety of different doses of MB07133

SUMMARY:
A randomized, open, multicenter clinical trial design was adopted, planned to be conducted in three stages, with 91 participants expected to be included in the study to evaluate the efficacy, tolerance, and safety of different doses of MB07133 in the treatment of unresectable advanced primary liver cancer.

DETAILED DESCRIPTION:
first stage：The investigators plan to recruit 20 cases for mid dose group exploration: the injection MB07133600mg/m2/day group and the 1200mg/m2/day group, with 10 cases recruited for each group. The treatment cycle is 28 days, with each dose group receiving 7 days of medication and 21 days of rest per cycle.

second stage：Based on the data results of the first stage, the 1200mg/m2/day dose group MB07133 was selected for further expansion, with the same administration method as the first stage. Plan to recruit 30 subjects.

third stage：Based on the treatment results of H201110LC3, the 1800mg/m2/day dose group was selected for further expansion, and 40 subjects were recruited with the same administration method as the first stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 75 years old (including 18 and 75 years old), regardless of gender;
2. Patients with advanced unresectable hepatocellular carcinoma confirmed by pathological diagnosis (pathological tissue/cytology) or clinical diagnosis (dynamic enhanced MRI/dynamic enhanced CT scan), who have failed first-line treatment or lack/do not have first-line standard treatment conditions;
3. At least one measurable lesion in the liver (in accordance with RECIST version 1.1 standard);
4. Child-Pugh liver function score: A/B (≤ 7 points);
5. Expected survival time ≥ 12 weeks;
6. ECOG score of 0 or 1;
7. Patients who have completed chemotherapy/radiation therapy for tumors for at least 4 weeks (those who have received chemotherapy with nitrosoureas and mitomycin for at least 6 weeks, those who have received small molecule targeted drugs (sorafenib, lovatinib) for at least 2 weeks), or those who have received chemotherapy/radiation therapy for at least 5 half-lives (the time limit shall be the longer); Surgical treatment>4 weeks, and the end time of the last intervention, radiotherapy, and ablation treatment>4 weeks;
8. Not using any anti-tumor drugs within 2 weeks before the first medication (including but not limited to the following modern Chinese medicine preparations with indications for liver cancer: Delisheng injection, Kanglaite injection or soft capsules, Aidi or Kangsaidi injection, elemene, Huaier granules, and Ganfule tablets);
9. Active hepatitis B patients should be controlled accordingly, and continue to take antiviral drugs and monitor liver function and hepatitis B virus load (for example, HBV DNA>104 copies/ml (2000IU/ml), and take antiviral drugs at least one week before use, and the virus quantity shows a downward trend);
10. If the main organs function normally, they meet the following standards:A. Blood routine examination: HGB ≥ 90 g/L; ANC ≥ 1.5 × 109/L; PLT ≥ 80 × 109/L;B. Biochemical examination: ALB ≥ 28 g/L; ALT and AST ≤ 5.0 × ULN; TBIL ≤ 1.5 × ULN; Creatinine ≤ 1.5 × ULN; The electrolyte is normal or normal after treatment or judged by the researcher to be abnormal without clinical significance;C. Urinary routine examination: Urinary protein ≤ 1+, such as urinary protein 2+, but 24-hour urinary protein<1.0g can be included in the group;. ECG results: QTcB<470ms for males and<480ms for females;
11. Those who agree to use effective non pharmacological contraceptive measures during the trial period;
12. The patient voluntarily signs a written informed consent form.

Exclusion Criteria:

1. Moderate or higher amounts of chest/ascites with clinical symptoms; Those who have received chest/ascites drainage within the past month; Only a small amount of chest/ascites found on imaging without symptoms can be included in the group;
2. Previous history of liver transplantation;
3. Obstructive jaundice and liver failure, resulting in hepatic encephalopathy; Tumor invading the inferior vena cava and forming a tumor thrombus in the inferior vena cava; If histological/pathological results can be provided, those with fibrous lamellar or sarcomatoid types cannot be included in the group;
4. Patients with other primary malignant tumors within 5 years, except for non melanoma skin cancer and cervical cancer in situ that have received sufficient treatment;
5. Individuals with active bleeding or abnormal coagulation function (PT>16s, APTT>43s, INR ≥ 2), bleeding tendency, or undergoing thrombolysis, anticoagulation, or antiplatelet therapy (except for those who require heparin due to PICC or deep venous catheterization); Those with significant bleeding/loss of blood (greater than 450ml) within 28 days;
6. Simultaneously taking drugs (such as amiodarone, quinidine, etc.) that may prolong QTc and/or induce torsade de pointe (Tdp);
7. Pregnant or lactating women;
8. Any significant clinical and laboratory abnormalities that the researchers think affect the safety evaluation, such as: serious or medically important infections, uncontrolled diabetes (glycosylated hemoglobin>9%), patients with hypertension who cannot be reduced to the following range after treatment with two or less antihypertensive drugs (systolic pressure<160 mmHg, diastolic pressure<100 mmHg), peripheral neuropathy of grade II or above (CTC AE V5.0) Congestive heart failure, myocardial infarction within 6 months, etc;
9. Patients with unstable brain metastasis, meningeal metastasis, and mental disorders; Patients with stable brain metastasis after treatment (no need for treatment for at least 4 weeks) can be enrolled in the group;
10. Have a history of gastrointestinal bleeding within 3 months in the past or have a clear tendency for gastrointestinal bleeding, such as those who are known to have local active ulcer lesions or have positive fecal occult blood and continue to be positive after retesting for 3 days;
11. Patients with significantly abnormal glomerular filtration rate (creatinine clearance rate ≤ 60ml/min, calculated according to the CKD-EPI formula, see Appendix 19.2);
12. Active hepatitis C, that is, those who are anti HCV positive and HCV RNA positive, and those who turn negative for HCV RNA after treatment can be included in the group;
13. HIV antibody positive individuals; Treponema pallidum antibody positive;
14. Those who use any drug or substance known to strongly inhibit or induce CYP3A4 liver microsomal enzyme 28 days prior to the use of the study drug (see the section on prohibited drugs for details);
15. Subjects suspected to have a history of allergy to araC or similar drugs;
16. Symptoms of gout and blood uric acid>430umol/L;
17. Any known deficiency in glutathione metabolism or the need for high doses of acetaminophen/Tylenol ® (>1 g/day), or subjects who require or use medication doses that will consume glutathione;
18. Patients who are unable to undergo enhanced magnetic resonance imaging, such as those who are allergic to magnetic resonance imaging agents, those who have a heart pacemaker, aneurysm surgery, or those who have metal objects such as steel nails and plates in their bodies; Women with an intrauterine device (IUD) need to consider the situation;
19. Patients who have participated in clinical trials of other drugs and used the study drug within 28 days prior to the use of the study drug (calculated based on the last use of the study drug);
20. Subjects who the researchers believe have other factors that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Screening period, every 2 cycles after treatment（each cycle is 28 days）until the date of first documented progression or date of death from any cause（No more than 24 cycles are expected）.
  The time between the first medication and the occurrence (progression) or (death) of the tumor (for any reason).

SECONDARY OUTCOMES:
OS | Treatment period and follow-up period until the date of death from any cause（Up to 24 months after the last subject was enrolled）.
  The time between the first medication use and (for any reason) death
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From the beginning of medication to 35 days after the last administration
  Adverse events occurring after treatment, as well as laboratory tests, vital signs, and electrocardiogram

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China